CLINICAL TRIAL: NCT03474835
Title: Ischemic Heart Disease in Male With Prostate Adenocarcinoma: Clinical and Pathogenetic Aspects of Diagnostics, Prognosis and Treatment
Brief Title: Ischemic Heart Disease in Male With Prostate Adenocarcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dnipropetrovsk State Medical Academy (Other)
Responsible Party: Principal Investigator, Oksana Sirenko, professor assistant, Dnipropetrovsk State Medical Academy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 832/18
Record Dates: First submitted 2018-02-28; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Ischemic Heart Disease; Prostate Adenocarcinoma
Keywords: atherosclerosis; angiogenesis; cardiooncology
MeSH Terms: conditions — Myocardial Ischemia; Atherosclerosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ISCHEMIC HEART DISEASE and PROSTATE ADENOCARCINOMA (Other)
  Interventions: Diagnostic Test: ISCHEMIC HEART DISEASE diagnostic
- ISCHEMIC HEART DISEASE and PROSTATE hyperplasia (No Intervention)

INTERVENTIONS:
Diagnostic Test: ISCHEMIC HEART DISEASE diagnostic — ISCHEMIC HEART DISEASE diagnostic
  Arms: ISCHEMIC HEART DISEASE and PROSTATE ADENOCARCINOMA

SUMMARY:
The purpose of the study: to increase the efficiency of diagnosis, treatment and prediction of the course of coronary heart disease in patients with adenocarcinoma of the prostate gland, depending on the hormonal status by determining the cardiovascular risk factors, factors of angiogenesis, structural and functional state of the heart, coronary vessels, kidney damage and their pharmacological correction.

DETAILED DESCRIPTION:
Research methods:

1. general-clinical examination
2. Laboratory methods:

   * estimation of the generally accepted laboratory parameters
   * determination of blood lipid profile
   * Determination of the level of highly sensitive CRP by the method of immuno-enzyme analysis,
   * determination of the level of proteinuria, creatinine by the method of immuno-enzyme analysis with the subsequent calculation of GFR
   * determination of the level of insulin by the method of immuno-enzyme analysis with the subsequent calculation of indices of insulin resistance,
   * determination of the level of blood testosterone by the method of immuno-enzyme analysis,
   * determination of the levels of vascular-endothelial growth factor, angiosetamine by the immuno-enzyme assay,
3. Echo-doppler examination of vessels (endothelium-dependent vasodilatation with reactive hyperemia, determination of the thickness of CIM, GPI)
4. Ultrasound examination of the main vessels of the head and neck
5. ECG
6. Daily monitoring of BP
7. CT-angiographic examination of coronary vessels with the definition of the index of calcification
8. Statistical methods

ELIGIBILITY:
Inclusion Criteria:

* men aged 45-75 years
* presence of verified diagnosis of adenocarcinoma of the prostate gland,
* stable antitumor therapy for 6 months, verified diagnosis of CAD,
* stable cardiological therapy for the past 3 months,
* voluntary informed consent to participate in the study.

Exclusion Criteria:

* age older than 75 years,
* female sex,
* metastatic lesion,
* chronic heart failure of the III-IV functional class (FC),
* arrhythmias that cause hemodynamic impairment and require antiarrhythmic correction (including ventricular arrhythmias of high gradation, atrial flutter , paroxysmal tachycardia, sinus node weakness syndrome, 2-3-degree AV block),
* AMI, acute cerebrovascular accident,
* diabetes mellitus (insulin-dependent diabetes mellitus) with a level of NvA1s> 7%, hyperthyroidism and hypothyroidism level of TSH> 10 mD / L, chronic renal failure (GFR <30 ml / min / 1.73 m2),
* acute cardiac and renal insufficiency,
* obesity 4 degrees,
* cachexia.

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-04-15 (Estimated); Study Completion 2019-01-15 (Estimated)

PRIMARY OUTCOMES:
cardiovascular events | 1 year
  cardiovascular events development - myocardial infarction, stroke

CONTACTS AND LOCATIONS:
Locations (1):
- SE Dnipropetrovsk medical academy, Dnipro, Ukraine